CLINICAL TRIAL: NCT05688072
Title: Trunk Oriented Exercises Versus Whole-body Vibration on Abdominal Thickness and Balance in Children With Duchenne Muscular Dystrophy
Brief Title: Trunk Oriented Exercises Versus Whole-body Vibration for Duchenne Muscular Dystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Shafiek Mustafa Saleh, assistance professor doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Treatment of Duchenne syndrome
Record Dates: First submitted 2023-01-08; First posted 2023-01-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Muscular Dystrophy, Duchenne Type
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (A) (Active Comparator)
  Interventions: Other: trunk oriented exercise
- Study group (B) (Active Comparator)
  Interventions: Other: whole body vibration

INTERVENTIONS:
Other: trunk oriented exercise — trunk oriented exercises include: stretching exercises, stabilization exercises (active or active-assisted), arm exercises in fixed trunk position, trunk-oriented exercises (active or active-assisted), trunk mobilization (sitting and lying position), and functional reaching exercises with different ranges of motion in shoulder elevation
  Arms: study group (A)
Other: whole body vibration — WBV application technique. The children assume a full squatting position on a vibration platform. The apparatus will set at a frequency of 30 Hz, an amplitude of 2 mm, and a duration of 5 min. The children were instructed to remain in squatting position after the vibration started and to report any discomfort that arose. At the end of 5 min, the vibration turned off automatically. Thereafter, the children rested for 1 min. They were then asked to stand on the vibration platform while supported by the therapist for 5 min, with the same parameters as those used in the squatting position. The total time of application of WBV in each session was 10 min.
  Arms: Study group (B)

SUMMARY:
The abdominal muscles play an important role in stabilizing the trunk and providing postural stability. Children with Duchene muscular dystrophy have weak muscles, which may impair postural adjustments. These postural adjustments are required for gait and dynamic balance during the daily living activities.

ELIGIBILITY:
Inclusion criteria:

* diagnosed as Duchenne muscular dystrophy,
* aged from 6 to 10 years,
* having grade 3+ muscle strength in lower limbs and trunk muscles.
* had functional range of motion for upper and lower limb joints,
* able to walk alone level I and II of Ambulation function classification system for DMD (AFCSD)
* Exclusion criteria:
* congenital or acquired skeletal deformities or cardiopulmonary dysfunction,
* had undergone previous orthopedic surgery in lower limbs,
* had abnormal motor development or neurological disease that affect balance
* and gait, and
* behavioral problems causing inability to cooperate during the study.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
abdominal muscle thickness | change from base line at 4 weeks.
  The thickness of four abdominal muscles will be measured with ultrasonography (device type GE Logiq P6) with a frequency of 7.5 MHz. The probe will be placed 2 or 3 cm from the midline, using the umbilicus as a landmark, then will be moved in a semi-circular motion until the deepest image on the screen, the TA, will be visible. To confirm this position and measure the thickness, a skin marker pen will be used. The probe will be then moved in an oblique manner to detect the thickness of the EO, IO, RA, and TA. A large amount of contact gel will be used, and the probe pressure will be adjusted to obtain optimal values of muscle thickness. After image capture, a vertical line will drawn between the superficial and deep aponeurosis to determine muscle thickness.

SECONDARY OUTCOMES:
balance assessment | change from base line at 4 weeks.
  the Biodex Balance System (BBS) (Biodex medical system, Shirley, New York) will be used for balance assessment.
  Before the evaluation procedures all children will be given an explanatory session to be aware about the different test steps, also the support rails and biofeedback display screen will be adjusted for each child to ensure comfort and safety during the test procedure, then each child will be trained 1 min for adaptation to the machine. During the test, children will be instructed to stand on the platform in the most comfortable posture, and maintain their visual level by focusing straight ahead on the monitor. The platform will be unlocked and children will be allowed to adjust their foot placement until a comfortable standing position will be achieved while they simultaneously maintained a moving pointer at the center point on the monitor and children will be encouraged to maintain the moving pointer at the center point throughout the test.

CONTACTS AND LOCATIONS:
Locations (1):
- marwa S saleh, Giza, Egypt

REFERENCES:
- [Derived] Ali MS, Saleh MS. Trunk-oriented Exercises Versus Whole-body Vibration on Abdominal Thickness and Balance in Children with Duchene Muscular Dystrophy. J Musculoskelet Neuronal Interact. 2024 Mar 1;24(1):47-54. PMID 38427368